CLINICAL TRIAL: NCT01851824
Title: A PHASE I, OPEN-LABEL, MULTICENTER, 3-PERIOD, FIXED-SEQUENCE STUDY TO INVESTIGATE THE EFFECT OF VEMURAFENIB ON THE PHARMACOKINETICS OF A SINGLE ORAL DOSE OF ACENOCOUMAROL IN PATIENTS WITH BRAFV600 MUTATION-POSITIVE METASTATIC MALIGNANCY
Brief Title: A Study of the Effect of Vemurafenib on the Pharmacokinetics of Acenocoumarol in Patients With BRAFV600 Mutation-Positive Metastatic Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GO28397; 2012-003706-27 (EudraCT Number)
Record Dates: First submitted 2013-05-03; First posted 2013-05-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Malignant Melanoma, Neoplasms
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Acenocoumarol; Vemurafenib

ARMS (1):
- Acenocoumarol + Vemurafenib (Experimental)
  Interventions: Drug: acenocoumarol; Drug: vemurafenib

INTERVENTIONS:
Drug: acenocoumarol — 4 mg single oral doses on Days 1 and 23
Drug: vemurafenib — 960 mg orally bid, 20 days (Days 4-23)
  Other Names: Zelboraf

SUMMARY:
This open-label, multicenter, 3-period, fixed-sequence study will evaluate the effect of multiple doses of vemurafenib on the pharmacokinetics of a single dose of acenocoumarol in participants with BRAFV600 mutation-positive metastatic malignancies. Participants will receive a single dose of acenocoumarol 4 mg orally on Day 1 and Day 23, vemurafenib 960 mg orally twice daily on Days 4-26. After completion of pharmacokinetic assessments on Day 26, eligible participants will have the option to continue treatment with vemurafenib as part of an extension study (GO28399 [NCT01739764]).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-70 years of age
* Patients with either unresectable Stage IIIc or IV BRAFV600 mutation-positive metastatic melanoma or other malignant BRAFV600 mutation-positive tumor type and who have no acceptable standard treatment options
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Full recovery from any major surgery or significant traumatic injury at least 14 days prior to the first dose of study treatment
* Adequate hematologic and end organ function
* Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to use 2 effective methods of contraception as defined by protocol during the course of the study and for at least 6 months after completion of study treatment

Exclusion Criteria:

* Prior treatment with vemurafenib or other BRAF inhibitor within 42 days of Day 1
* Prior anti-cancer therapy within 28 days (6 weeks for nitrosureas or mitocyn C, or 14 days for hormonal therapy or kinase inhibitors) before the first dose of study treatment Day 1
* Palliative radiotherapy within 2 weeks prior to first dose of study treatment Day 1
* Experimental therapy within 4 weeks prior to first dose of study treatment Day 1
* History of clinically significant cardiac or pulmonary dysfunction, including current uncontrolled Grade >/=2 hypertension or unstable angina
* Current Grade >/=2 dyspnea or hypoxia or need for oxygen supplementation
* History of myocardial infarction within 6 months prior to first dose of study treatment
* Active central nervous system lesions (i.e. participants with radiographically unstable, symptomatic lesions)
* History of bleeding or coagulation disorders
* Allergy or hypersensitivity to vemurafenib or acenocoumarol formulations
* History of malabsorption or other condition that would interfere with the enteral absorption of study treatment
* Participants with VKORC1 mutations (1639G→A, 1173C→T) in either one allele (heterozygous)or two alleles (homozygous)
* Participants with CYP2C9*3 mutations in either one allele (heterozygous) or two alleles (homozygous)
* History of clinically significant liver disease (including cirrhosis), current alcohol abuse, or active hepatitis B or hepatitis C virus infection
* Human immunodeficiency virus (HIV) infection requiring antiretroviral treatment, or AIDS-related illness
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single-dose acenocoumarol under conditions of vemurafenib steady-state exposure: Area under the concentration-time curve (AUC) | Pre-dose and up to 72 hours post-dose
Pharmacokinetics of single-dose acenocoumarol under conditions of vemurafenib steady-state exposure: Maximum plasma concentration (Cmax) | Pre-dose and up to 72 hours post-dose
Pharmacokinetics of single-dose acenocoumarol under conditions of vemurafenib steady-state exposure: Time to maximum plasma concentration (Tmax) | Pre-dose and up to 72 hours post-dose
Pharmacokinetics of single-dose acenocoumarol under conditions of vemurafenib steady-state exposure: Terminal half-life (t1/2) | Pre-dose and up to 72 hours post-dose
Pharmacokinetics of single-dose acenocoumarol under conditions of vemurafenib steady-state exposure: Apparent clearance (CL/F) | Pre-dose and up to 72 hours post-dose

SECONDARY OUTCOMES:
Safety: Incidence of Adverse Events and Serious Adverse Events | approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Wodonga, New South Wales, Australia
- Germany (3):
  - Buxtehude
  - Essen
  - Mannheim
- Greece (2):
  - Crete
  - Thessaloniki
- Budapest, Hungary
- Netherlands (3):
  - Amsterdam
  - Maastricht
  - Utrecht
- New Zealand (2):
  - Auckland
  - Christchurch
- Portugal (2):
  - Lisbon
  - Porto
- Belgrade, Serbia
- Spain (2):
  - Barcelona, Barcelona
  - Madrid, Madrid